CLINICAL TRIAL: NCT06503094
Title: The Safety and Efficacy of CD19 & CD20 Bispecific CAR T Cells in Treating Relapsed / Refractory B Cell Hematological Tumors
Brief Title: CD19 & CD20 Bispecific CAR T Cells for Relapsed / Refractory B Cell Hematological Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Hebei Taihe Chunyu Biotechnology Co., Ltd (Industry); Zhujiang Hospital (Other); Jingzhou Central Hospital (Other); Shiyan People's Hospital (Unknown); Xiangyang Central Hospital (Other); Yichang Central People's Hospital (Other)
Responsible Party: Principal Investigator, MEI HENG, : Proferssor, Cheif Doctor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19 & CD20 bispecific CAR T
Record Dates: First submitted 2024-06-17; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: B-Cell Lymphoblastic Leukemia/Lymphoma
Keywords: CAR-T; dual-target; Relapsed / Refractory B Cell Hematological Tumors
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effective of CD19&CD20 bispecific CAR-T cells (Experimental): The infusion dose range of cells in this trial is recommended: 2 to 6 10^6 And CAR-T cells / kg.
  Interventions: Drug: CD19&CD20 bispecific CAR-T cells

INTERVENTIONS:
Drug: CD19&CD20 bispecific CAR-T cells — Each patient will receive CD19&CD20 bispecificCAR-T cells by intravenous infusion on day 0.

SUMMARY:
This study is a multi-center, open, prospective single-arm clinical study of patients with relapsed / refractory B cell hematological tumors to evaluate the safety and efficacy of CD19 & CD20 bispecific CAR-T cells in relapsed / refractory B cell hematological tumors while collecting pharmacokinetics and pharmacodynamics indicators of CAR-T cells.

DETAILED DESCRIPTION:
Since 2010, CAR-T ( chimeric antigen receptor T cell) therapy has shown good results in tumor treatment and has achieved positive clinical therapeutic effects in hematological tumors. The structure of the dual-target CAR-T of CD19 & CD20 is designed with a 4-1BB costimulatory domain and an antigenic recognition region with a tandem structural sequence to recognize CD20 or CD19 by a single structure. CD19 & CD20 bispecific CAR-T cells can identify CD 19 or CD 20 with the advantage that the single target CAR-T does not have, reducing the possibility of target loss. The structure has been optimized to enhance the safety to treat B cell-derived hematological tumors (at least CD19 positive or CD20 positive).

ELIGIBILITY:
Inclusion Criteria:

* Fully understand and voluntarily sign the informed consent form, and be willing and able to comply with the visit, treatment protocol, laboratory tests, and other study requirements specified in the flow sheet;
* CD 19 + / CD 20 + B cell hematological tumor was confirmed by pathological and histological examination, and the patient met the following criteria for relapsed or refractory B cell hematological tumor:

  1. Refractory / relapsed B lymphocytic leukemia (1 of the following 4 items can be met):

     i . Recurrence within 6 months of first remission; ii. Primary refractory without complete remission after 2 cycles of standard chemotherapy regimen; iii. No complete remission or recurrence after first-line or multiline salvage chemotherapy; iv. Not eligible for HSCT conditions, abandonment of HSCT, or relapse after HSCT due to conditional limitations.
  2. Refractory / relapsed B-cell lymphoma (meet the following item 1 of the first 4 items plus item 5):

i . After four courses of chemotherapy with a standard regimen, tumor shrinkage was less than 50% or disease progression; ii . CR after standard regimen chemotherapy, but relapsed within 6 months; iii.2 or more recurrences after CR; iv . Not suitable for hematopoietic stem cell transplantation, or abandoning HSCT due to conditional restrictions or relapse after hematopoietic stem cell transplantation; v . Subject must have received prior adequate treatment, including at least: a monoclonal antibody against CD 20 and combination chemotherapy containing an anthracycline drug agent.

* B-cell hematological tumors include the following 3 categories:

  1. B-cell acute lymphoblastic leukemia (B-ALL);
  2. Indolent B-cell lymphoma (CLL, FL, MZL, LPL, HCL);
  3. Invasive B-cell lymphoma (DLBCL, BL, and MCL);
* With measurable or evaluable lesions: Lymphoma patients require a single lesion 15mm or 2 or more lesions 10mm; patients with leukemia require persistent positive or positive recurrence of bone marrow MRD.
* Subjects with the Eastern Cooperative Oncology Group (ECOG) fitness scores of 0 to 2.
* The results of FCM or immunohistochemical detection of tumor antigen (CD 19 / CD 20) were positive.
* The estimated survival period is more than 3 months starting from the signing of the informed consent form.

Exclusion Criteria:

* Appearance of one of the following cardiac criteria: atrial fibrillation; myocardial infarction in the last 12 months; prolonged QT syndrome or secondary QT extension, as judged by the investigator. Echocardiography LVSF <30% or LVEF <50%; clinically significant pericardial effusion; cardiac insufficiency NYHA (New York Heart Association) III or IV (confirmed by echocardiography within 12 months of treatment).
* Active GVHD.
* History of severe pulmonary function impairment disease.
* Other malignant tumors in the advanced stage.
* Severe infection or persistent infection that cannot be effectively controlled.
* Combined with severe autoimmune disease or innate immune deficiency.
* Active hepatitis (hepatitis B virus deoxyribonucleic acid [HBV-DNA 500 IU / ml and abnormal liver function] or hepatitis C antibody [HCV-Ab] positive, HCV-RNA above the lower limit of detection of the analytical method and abnormal liver function).
* Human immunodeficiency virus (HIV) infection or syphilis infection.
* History of severe allergies to biological products (including antibiotics).
* There are central nervous system disorders, such as uncontrolled epilepsy, cerebrovascular ischemia/hemorrhage, dementia, cerebellar diseases, etc..
* Female patients are in pregnancy and lactation, or have a pregnancy plan within 12 months.
* situations where the investigator may increase the risk or interfere with the test results.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-14 (Actual); Primary Completion 2025-12-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) of administering CD19&CD20 dual-target CAR-T cells In the treatment of relapsed/refractory B-cell hematologic tumors | within 3 years after infusion
  Disease overall response rate (ORR) will be assessed from CAR-T cell infusion to death or last follow-up (censored).
Incidence of Treatment-related Adverse Events | within 3 years after infusion
  Therapy-related adverse events (AE), including severe adverse events (SAE) and laboratory outliers with clinical significance, will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).
Complete response rate (CR) of administering CD19&CD20 dual-target CAR-T cells In the treatment of relapsed/refractory B-cell hematologic tumors | within 3 years after infusion
  CR will be assessed from CAR-T cell infusion to death or last follow-up (censored).
Partial response rate (PR) of administering CD19&CD20 dual-target CAR-T cells In the treatment of relapsed/refractory B-cell hematologic tumors | within 3 year after infusion
  PR will be assessed from CAR-T cell infusion to death or last follow-up.

SECONDARY OUTCOMES:
Overall survival (OS) of administering CD19&CD20 dual-target CAR-T cells in the treatment of relapsed/refractory B-cell hematologic tumors | within 3 years after infusion
  OS will be assessed from CAR-T cell infusion to death or last follow-up (censored).
Progress-free survival (PFS) of administering CD19&CD20 dual-target CAR-T cells in the treatment of relapsed/refractory B-cell hematologic tumors | within 3 years after infusion
  PFS will be assessed from CAR-T cell infusion to death or last follow-up (censored).
Event-free survival (EFS) of administering CD19&CD20 dual-target CAR-T cells in the treatment of relapsed/refractory B-cell hematologic tumors | within 3 years after infusion
  EFS will be assessed from CAR-T cell infusion to death or last follow-up (censored).

OTHER OUTCOMES:
In vivo expansion and survival of CD19&CD20 dual-target CAR-T cell therapy in relapsed/refractory B-cell hematological malignancies | within 3 years after infusion
  Quantity of CAR-T-CD19 CAR copies in bone marrow, peripheral blood and cerebrospinal fluid will be determined by using flow cytometry and quantitative polymerase chain reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Heng, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Background] Lee DW, Kochenderfer JN, Stetler-Stevenson M, Cui YK, Delbrook C, Feldman SA, Fry TJ, Orentas R, Sabatino M, Shah NN, Steinberg SM, Stroncek D, Tschernia N, Yuan C, Zhang H, Zhang L, Rosenberg SA, Wayne AS, Mackall CL. T cells expressing CD19 chimeric antigen receptors for acute lymphoblastic leukaemia in children and young adults: a phase 1 dose-escalation trial. Lancet. 2015 Feb 7;385(9967):517-528. doi: 10.1016/S0140-6736(14)61403-3. Epub 2014 Oct 13. PMID 25319501
- [Background] Ali SA, Shi V, Maric I, Wang M, Stroncek DF, Rose JJ, Brudno JN, Stetler-Stevenson M, Feldman SA, Hansen BG, Fellowes VS, Hakim FT, Gress RE, Kochenderfer JN. T cells expressing an anti-B-cell maturation antigen chimeric antigen receptor cause remissions of multiple myeloma. Blood. 2016 Sep 29;128(13):1688-700. doi: 10.1182/blood-2016-04-711903. Epub 2016 Jul 13. PMID 27412889
- [Background] Khalil DN, Smith EL, Brentjens RJ, Wolchok JD. The future of cancer treatment: immunomodulation, CARs and combination immunotherapy. Nat Rev Clin Oncol. 2016 May;13(5):273-90. doi: 10.1038/nrclinonc.2016.25. Epub 2016 Mar 15. PMID 26977780
- [Background] Maude SL, Frey N, Shaw PA, Aplenc R, Barrett DM, Bunin NJ, Chew A, Gonzalez VE, Zheng Z, Lacey SF, Mahnke YD, Melenhorst JJ, Rheingold SR, Shen A, Teachey DT, Levine BL, June CH, Porter DL, Grupp SA. Chimeric antigen receptor T cells for sustained remissions in leukemia. N Engl J Med. 2014 Oct 16;371(16):1507-17. doi: 10.1056/NEJMoa1407222. PMID 25317870
- [Result] Cohen AD, Garfall AL, Stadtmauer EA, Melenhorst JJ, Lacey SF, Lancaster E, Vogl DT, Weiss BM, Dengel K, Nelson A, Plesa G, Chen F, Davis MM, Hwang WT, Young RM, Brogdon JL, Isaacs R, Pruteanu-Malinici I, Siegel DL, Levine BL, June CH, Milone MC. B cell maturation antigen-specific CAR T cells are clinically active in multiple myeloma. J Clin Invest. 2019 Mar 21;129(6):2210-2221. doi: 10.1172/JCI126397. PMID 30896447